CLINICAL TRIAL: NCT05223543
Title: The Presence of N-Methyl-D-Aspartic Acid Receptor (NMDA-R) Antibodies in Serums of Women With Pathology Proven Dermoid Cyst and Examining the Relationship of Cyst Characteristics
Brief Title: Paraneoplastic Neurologic Encephalitis and Mature Cystic Teratoma
Acronym: dermoid_cyst
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Noam Smorgick MD, Director of Minimally Invasive Gynecology, Assaf-Harofeh Medical Center
Other Study IDs: 0194-18; 0194-18 (Other: Shamir medical center)
Record Dates: First submitted 2021-09-12; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Ovarian Dermoid Cyst
MeSH Terms: conditions — Teratoma, Ovarian | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples with extraction of plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood sample — extraction of blood samples from women undergoing ovarian cystectomy or oophorectomy due to suspected Dermoid cyst and analysing plasma for antibodies

SUMMARY:
Ovarian dermoid cyst, also known as benign mature teratoma, originate from germ cells in the ovary, and is the most common benign ovarian tumor (44-70%). Several reports documented a secretion of NMDA receptor antibodies from dermoid cyst. This receptor is found in different areas in the central nerves system (CNS) and the presence of plasma antibodies has been shown as a rare cause of neurologic presentation term paraneoplastic neurologic syndrome, which can be characterized by mood disorder, psychiatric and neurologic symptoms. In several case reports on young women, first presented with nonspecific neurologic symptoms, then followed by rapid deterioration of conscious, seizures and the need for ventilation support, ovarian teratoma was diagnosed. In 2007 an association between N-Methyl-D-Aspartic acid (NMDA) receptor antibody and encephalitis was first described. More than 50% of paraneoplastic encephalitis were related to teratomas, most often from an ovarian origin. Therapy includes tumor resection, steroids, plasmapheresis and immunosuppressive drugs. The investigators recently published a retrospective cohort study analyzing 233 patients who were operated in their institution with pathology proven dermoid. In this study 2 patients presented with paraneoplastic syndrome (0.85%). No prospective study has been published to date to examine the association between antibody titer and dermoid cyst characteristics and the paraneoplastic phenomenon. The investigators wish to conduct a prospective study in which plasma samples will be obtained from patients asymptomatic for neurologic or psychiatric symptoms, undergoing surgery for ovarian dermoid cyst, due to gynecology indication (e.g size, symptoms) in order to identify antibodies against CNS NMDA-R in their plasma prior to cyst removal. If NMDA receptor antibodies will be discovered in asymptomatic patients it may be prudent to examine all serums of women who are diagnosed with ovarian mature teratoma, and offer a surgical removal in order to prevent a possible neurologic sequela in the presence of these antibodies.

DETAILED DESCRIPTION:
The data is collected by examining women's serum for the presence of NMDA-R antibodies, using special ELISA (enzyme-linked immunoabsorbent assay) kits. The analysis will be made by Dyn diagnostics labs. The investigators will obtain a blood sample prior to the operation for cystectomy or oophorectomy and after a written informed consent by the patient. All specimen are sent to pathology examination and only proven dermoid cyst will eventually be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Women admitted for surgery for removal of suspected dermoid cysts
2. No neurologic symptoms

Exclusion Criteria:

1. No surgical specimen available
2. The cyst pathology does not show dermoid cyst characteristics

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women in reproductive years
Study Population: women in reproductive years undergoing cystectomy or oopherectomy due to suspected ovarian dermoid cyst
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
prevalence of NMDA receptor antibodies | baseline, pre-surgery
  to identify the prevalence of antibodies and titer in the presence of ovarian dermoid cyst in neurology asymptomatic patients

CONTACTS AND LOCATIONS:
Overall Officials: Noam Smorgick, M.D, Study Director — Assaf-Harofeh Medical Center
Locations (1):
- Shamir medical center, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ayhan A, Bukulmez O, Genc C, Karamursel BS, Ayhan A. Mature cystic teratomas of the ovary: case series from one institution over 34 years. Eur J Obstet Gynecol Reprod Biol. 2000 Feb;88(2):153-7. doi: 10.1016/s0301-2115(99)00141-4. PMID 10690674
- [Background] Dalmau J, Gleichman AJ, Hughes EG, Rossi JE, Peng X, Lai M, Dessain SK, Rosenfeld MR, Balice-Gordon R, Lynch DR. Anti-NMDA-receptor encephalitis: case series and analysis of the effects of antibodies. Lancet Neurol. 2008 Dec;7(12):1091-8. doi: 10.1016/S1474-4422(08)70224-2. Epub 2008 Oct 11. PMID 18851928
- [Background] Vitaliani R, Mason W, Ances B, Zwerdling T, Jiang Z, Dalmau J. Paraneoplastic encephalitis, psychiatric symptoms, and hypoventilation in ovarian teratoma. Ann Neurol. 2005 Oct;58(4):594-604. doi: 10.1002/ana.20614. PMID 16178029
- [Background] Dalmau J, Tuzun E, Wu HY, Masjuan J, Rossi JE, Voloschin A, Baehring JM, Shimazaki H, Koide R, King D, Mason W, Sansing LH, Dichter MA, Rosenfeld MR, Lynch DR. Paraneoplastic anti-N-methyl-D-aspartate receptor encephalitis associated with ovarian teratoma. Ann Neurol. 2007 Jan;61(1):25-36. doi: 10.1002/ana.21050. PMID 17262855
- [Background] Li W, Jia D, Tong L, Lun Z, Li H. Anti-N-methyl-D-aspartate receptor encephalitis induced by bilateral ovarian teratomas with distinct histopathologic types: A case report and brief literature review. Medicine (Baltimore). 2019 Nov;98(48):e18148. doi: 10.1097/MD.0000000000018148. PMID 31770255
- [Result] Pekar-Zlotin M, Rabinovich I, Goldrat I, Vaknin Z, Gidoni Y, Zur-Naaman H, Maymon R, Smorgick N. Ovarian Dermoid Cysts Associated with Paraneoplastic Syndrome N-methyl-D-aspartic Acid Receptor Antibodies Encephalitis. J Minim Invasive Gynecol. 2021 Jun;28(6):1190-1193. doi: 10.1016/j.jmig.2020.09.018. Epub 2020 Sep 24. PMID 32979534